CLINICAL TRIAL: NCT03562117
Title: A Phase I, Open-Label, Single-Dose, Two-Part Study to Assess the Pharmacokinetics of Gepotidacin (GSK2140944) in Male and Female Adult Participants With Varying Degrees of Hepatic Impairment and in Matched Control Participants With Normal Hepatic Function
Brief Title: Pharmacokinetics (PK) Study of Gepotidacin (GSK2140944) in Adult Subjects With Varying Degrees of Hepatic Impairment and in Matched Control Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117352
Record Dates: First submitted 2018-05-15; First posted 2018-06-19 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Infections, Bacterial
Keywords: Child-Pugh classification; Open label; Hepatic Impairment; Gepotidacin
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Masking Description: There will be no masking, as this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Normal Hepatic function, Part 1 (Group D) (Experimental): The eligible subjects, with normal hepatic function, in this arm will receive a single oral dose of gepotidacin as 1500 milligram (mg), administered as 2 × 750 mg tablets on Day 1.
  Interventions: Drug: Gepotidacin
- Moderate hepatic impairment, Part 1 (Group B) (Experimental): The subjects in this arm, will be the one's with a Child-Pugh score of 7 to 9, and will receive a single oral dose of gepotidacin, as 1500 mg, administered as 2 × 750 mg tablets on Day 1.
  Interventions: Drug: Gepotidacin
- Mild hepatic impairment, Part 2 (Group A) (Experimental): The subjects in this arm, will be the one's with a Child-Pugh score of 5 to 6, and will receive a single oral dose of gepotidacin, as 1500 mg, administered as 2 × 750 mg tablets on Day 1. This will be optional arm.
  Interventions: Drug: Gepotidacin
- Severe hepatic impairment, Part 2 (Group C) (Experimental): The subjects in this arm, will be the one's, with a Child-Pugh score of 7 to 9, and will receive a single oral dose of gepotidacin, as 1500 mg, administered as 2 × 750 mg tablets, on Day 1.
  Interventions: Drug: Gepotidacin
- Normal Hepatic function, Part 2 (Group E) (Experimental): The eligible subjects, with normal hepatic function, will be matching with those enrolled in Part1, and will receive a single oral dose of gepotidacin as 1500 mg, administered as 2 × 750 mg tablets on Day 1.
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — It is an immediate-release tablet (1500 mg (2 x 750 mg), containing gepotidacin (free base) an inactive formulation excipients.

SUMMARY:
This is a two-part study which will evaluate the PK, safety, and tolerability of a single 1500 milligram (mg) oral dose of gepotidacin in subjects with normal hepatic function and in subjects with mild, moderate, and severe hepatic impairment. In Part 1, subjects with moderate hepatic impairment and subjects with normal hepatic function will be enrolled. Matching subjects with normal hepatic function in Part 1 (Group D), will be enrolled following the completion of all Day 3 assessments of the respective matched, hepatically impaired subject. In Part 2, subjects with mild (optional) and severe hepatic impairment and subjects with normal hepatic function will be enrolled concurrently based on the PK, safety, and tolerability data of Part 1. Subjects with mild hepatic impairment, may be studied if there is a significant difference in PK between subjects with moderate hepatic impairment and subjects with normal hepatic function. Subjects with severe hepatic impairment, will be studied in Part 2, provided that, the PK objectives are achieved in Part 1. A totals of 48 subjects, are planned to be enrolled in the study. The study duration is approximately of 44 days from Screening to Follow-up visit. The results from this study will enable the development of appropriate dosing recommendations in subjects with impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 80 years of age inclusive, at the time of signing the informed consent.
* Healthy subjects must be in clinically stable health as determined by the investigator based on medical history, clinical laboratory results (serum chemistry, hematology, urinalysis, and serology), vital sign measurements, 12-lead ECG results, and physical examination findings.
* Hepatically impaired subjects must have chronic (>6 months), stable (no acute episodes of illness within the previous 1 month prior to screening due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology. Subjects must also remain stable throughout the Screening period.
* Hepatically impaired subjects, will be classified, using the Child-Pugh classification system. Subjects must have, a Child-Pugh score, of 5 to 6 (mild hepatic impairment), 7 to 9 (moderate hepatic impairment), or 10 to 15 (severe hepatic impairment), with known medical history of liver disease (with or without a known history of alcohol abuse), and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, computed tomography scan, magnetic resonance imaging, or ultrasonography) associated with unambiguous medical history. If imaging study, or biopsy is not available, then the subject should have one of the following: Physical findings such as hepatomegaly, ascites, palmar erythema, spider angiomata, abdominal venous collaterals, gynecomastia, or other physical manifestations of hepatic disease Or Laboratory findings: ALT or AST elevation (> upper limit of normal [ULN]), alkaline phosphatase, or total bilirubin, or international normalized ratio (INR) elevation (>ULN) or an albumin value that is below the lower limit of normal laboratory reference range.
* Subjects with hepatic impairment may be taking medications, which in the opinion of the investigator, are believed to be therapeutic, and these medications should not interfere with the conduct of the study. Subjects with hepatic impairment should be on stable regimen of chronic medications for at least 7 days prior to dosing until completion of the Follow-Up Visit.
* Subjects with hepatic impairment must have platelet counts of 30,000 × 109/Liter of blood and have not had any major bleeding episodes within the past 6 months.
* Body weight >=45 kilogram (kg) and body mass index (BMI) within the range 18.5 to 40 kg/meter^2 (inclusive).
* Male subjects must agree to use contraception, as protocol from Day -1 until completion of the Follow-up Visit or, female subject will be eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applied Not a woman of childbearing potential (WOCBP) or A WOCBP who agrees to follow the contraceptive guidance from 30 days prior to study drug administration and until completion of the Follow-up Visit.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Subject has a clinically significant abnormality in past medical history or at the Screening physical examination (excluding hepatic insufficiency and other related medical conditions within the hepatically impaired populations, which should be stable for at least 1 month before study drug administration), that in the investigator's opinion, may place the subject at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current significant cardiac, renal, neurologic, gastrointestinal, respiratory, hematologic, or immunologic disease.
* Subject has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the subject at risk, in the opinion of the investigator.
* Female subject, has a positive pregnancy test result or is lactating at Screening or upon admission to the clinic.
* Subject has used a systemic antibiotic within 7 days of Screening.
* Subject has a confirmed history of Clostridium (C) difficile infection or a positive C. difficile toxin test, within 2 months before Screening.
* Subject has a history of drug and/or alcohol abuse within 6 months before Screening, as determined by the investigator, or subject has a positive drug screen at Screening or upon admission to the clinic. For subjects with hepatic impairment, and a positive drug screen result related to the use of prescription medications, is allowed per investigator review and approval, and tetrahydrocannabinol use is allowed per investigator review and approval.
* History of sensitivity to any of the study drugs, components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain intravenous cannula patency).
* Subject has used medications known to affect the elimination of serum creatinine (example (e.g); trimethoprim or cimetidine) or competitors of renal tubular secretion (e.g., probenecid) within 30 days before dosing.
* Subject must abstain from taking prescription or nonprescription drugs (including vitamins and dietary or herbal supplements), unless specified, within 7 days (or 14 days if the drug is a potential strong enzyme inducer) or 5 half-lives (whichever is longer) prior to study drug administration until completion of the Follow-Up Visit, unless, in the opinion of the investigator and Sponsor, the medication will not interfere with the study. Any exceptions (including subjects with hepatic impairment that will be on medications during the study), will be discussed with the sponsor or medical monitor on a case-by-case basis and the reasons will be documented.
* Previous exposure to gepotidacin, within 12 months prior to study drug administration.
* Subject has participated in a clinical trial and has received an investigational product within the following time period prior to study drug administration in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subject with normal hepatic function has presence of hepatitis B surface antigen or positive hepatitis C antibody test result at Screening or within 3 months prior to study drug administration. Subject with hepatic impairment has evidence of recent, acute infection with hepatitis B and/or hepatitis C within preceding 6 months. Hepatically impaired subjects with chronic hepatitis B or C (duration >6 months) will be eligible for enrolment.
* A positive test for human immunodeficiency virus antibody.
* Subject must be able to abstain from alcohol and limit use of nicotine and/or nicotine-containing products (up to 5 cigarettes/day is acceptable for subjects with hepatic impairment) for 24 hours before the start of dosing until after collection of the final PK sample. A positive alcohol or cotinine test is not exclusionary for subjects with hepatic impairment.
* Subject has clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at Screening or Day -1, other than those associated with underlying hepatic conditions or other stable medical conditions consistent with the disease process in subjects with hepatic impairment.
* Subject with normal hepatic function has a baseline corrected QT interval using the Fridericia formula (QTcF) of >450 milliseconds (msec) and subject with hepatic impairment has a baseline QTcF of >480 msec.
* Donation of blood in excess of 500 milliliter (mL) within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Subject is unable to comply with all study procedures, in the opinion of the investigator.
* Subject should not participate in the study, in the opinion of the investigator or Sponsor.
* Subjects with a pre-existing condition (except hepatic impairment) interfering with normal gastrointestinal (GI) anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of inflammatory bowel disease should be excluded. Subjects with a history of pepticulceration or pancreatitis within the preceding 6 months of screening, should be excluded.
* Subject with any previous GI surgery (except appendectomy or gall bladder removal >3 months prior to Screening) may be enrolled in this study only if, in the opinion of the investigator and the medical monitor, it is not expected to interfere with the study procedures or to pose an additional safety risk to the subject.
* Subject receiving lactulose who are medically unable to halt lactulose administration from 8 hours before dosing with study drug to 4 hours after dosing with study drug.
* Subjects with clinically active severe encephalopathy (grade 3 or 4) as judged by the investigator or significant central nervous system disease (e.g., dementia or seizures) which the investigator considers will interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject. Subjects with a prior history of severe encephalopathy, who are currently treated for this condition will receive the appropriate score for encephalopathy.
* Subjects with estimated creatinine clearance (Clcr) <=50 mL/minute (calculated by the Cockcroft-Gault Formula). If the result calculated by Cockcroft-Gault is between 40 and 50 mL/minute, then the site may complete a 24-hour urine collection to more specifically calculate the Clcr. A Clcr value <=50 mL/minute via 24-hour urine collection is also exclusionary.
* History of gastric or esophageal variceal bleeding within the past 6 months and for which varices have not been adequately treated with medication and/or surgical procedures.
* Subjects with electrolyte imbalance whose serum sodium levels are <=125 millimole per Liter (mmol/L); potassium levels are <=2.5 mmol/L; or calcium levels are <=6.1 mmol/L.
* Presence of hepatopulmonary or hepatorenal syndrome.
* Primary cholestatic liver diseases.
* History of liver transplantation or subjects in the severe hepatic impairment group that are expecting a liver transplant during the study participation period.
* Subjects with signs of active bacterial infection (including active spontaneous bacterial peritonitis).
* Subjects with transjugular intrahepatic portosystemic shunt placement within the past 3 months.
* Subjects with unstable cardiac function or subjects with hypertension whose blood pressure, that is not well controlled (based on the investigator's discretion).
* Diabetic subjects whose diabetes that is not controlled (based on the investigator's discretion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase I, non-randomized, open-label, parallel-group, multi-center, two-part study that evaluated the pharmacokinetics, safety, and tolerability of a single 1500 milligrams (mg) oral dose of gepotidacin in participants with normal hepatic function and in participants with mild, moderate, and severe hepatic impairment.
Pre-assignment Details: Twenty five participants were enrolled in the study. In part 1, normal hepatic function participants were matched to moderate hepatic impaired participants. In Part 2, participants with severe hepatic impairment were matched to normal hepatic function participants who participated in Part1.
Groups:
- Participants With Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of gepotidacin 1500 mg administered as 2 × 750 mg tablets on Day 1.
- Participants With Moderate Hepatic Impairment: Participants with moderate hepatic function having Child-Pugh score of 7 to 9 received a single oral dose of gepotidacin 1500 mg administered as 2 × 750 mg tablets on Day 1.
- Participants With Severe Hepatic Impairment: Participants with severe hepatic function having Child-Pugh score of 10 to 15 received a single oral dose of gepotidacin 1500 mg administered as 2 × 750 mg tablets on Day 1.
Period: Part 1, Up to 3 Days
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Started | 8 | 8 | 0
Completed | 7 | 8 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Part 2, Up to 3 Days
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Started | 8 (Only 1 additional participant with normal hepatic function enrolled in Part 2 received dosing) | 0 | 8
Completed | 8 | 0 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (5.70) | 62.5 (7.19) | 58.1 (6.15) | 60.1 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 8 | 7 | 8 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 1
  African American/African Heritage | 3 | 0 | 0 | 3
  White - White/Caucasian/European Heritage | 6 | 8 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero (Pre-dose) Extrapolated to Infinity (AUC[0-inf]) for Plasma Gepotidacin
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate pharmacokinetic (PK) parameters. PK parameter population consist of all participants in the PK Population, for whom valid and evaluable PK parameters were derived. This population was used in the assessment and characterization of PK parameters.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Hours*nanograms per milliliter | 15894.7 (44.1) | 19505.7 (42.6) | 25415.5 (30.1)

2. Primary Outcome: Maximum Observed Concentration (Cmax) for Plasma Gepotidacin
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Nanograms per milliliter | 3196.8 (85.0) | 3913.7 (64.1) | 5541.8 (42.7)

3. Secondary Outcome: AUC From Time 0 to the Time of the Last Quantifiable Concentration (AUC [0-t]) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Hours*nanograms per milliliter | 15512.9 (45.8) | 19151.6 (43.4) | 25066.8 (30.5)

4. Secondary Outcome: Time to First Occurrence (Tmax) of Cmax for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Hours | 3.000 [1.50 to 6.00] | 2.750 [2.50 to 4.00] | 2.250 [0.50 to 4.00]

5. Secondary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Hours | 0.50 [0.0 to 2.5] | 0.00 [0.0 to 1.0] | 0.00 [0.0 to 1.0]

6. Secondary Outcome: Apparent Oral Clearance (CL/F) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hours
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Liters per hours | 94.37 (44.1) | 76.90 (42.6) | 59.02 (30.1)

7. Secondary Outcome: Apparent Volume of Distribution of the Terminal Phase (Vz/F) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Liters | 1235.3 (57.5) | 944.7 (50.3) | 699.1 (41.7)

8. Secondary Outcome: Terminal-phase Rate Constant (Lambda_z) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Per hour | 0.07639 (14.9) | 0.08140 (12.3) | 0.08443 (15.2)

9. Secondary Outcome: Terminal Phase Half Life (t1/2) for Plasma Gepotidacin
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Hours | 9.073 (14.9) | 8.515 (12.3) | 8.210 (15.2)

10. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Single 12-lead ECG was obtained in a semi-supine position after 5 minutes rest using an ECG machine. Safety Population consists of all participants who received at least 1 dose of study drug and had at least one postdose safety assessment. Number of participants with abnormal-clinically significant and abnormal-not clinically significant values has been presented. Absolute QTc Interval >450 milliseconds (msec), absolute PR interval <110 msec and absolute QRS interval <75 msec was considered as clinically significant ECG findings.
Time Frame: 1.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post-dose
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Participants
  1.5 hours, not clinically significant | 1 | 6 | 3
  1.5 hours, clinically significant | 0 | 0 | 0
  2 hours, not clinically significant | 5 | 6 | 5
  2 hours, clinically significant | 0 | 0 | 0
  4 hours, not clinically significant | 6 | 6 | 5
  4 hours, clinically significant | 0 | 0 | 0
  8 hours, not clinically significant | 3 | 5 | 4
  8 hours, clinically significant | 0 | 0 | 0
  12 hours, not clinically significant | 2 | 4 | 2
  12 hours, clinically significant | 0 | 0 | 0
  24 hours, not clinically significant | 6 | 5 | 5
  24 hours, clinically significant | 0 | 0 | 0
  36 hours, not clinically significant | 2 | 5 | 4
  36 hours, clinically significant | 0 | 0 | 0
  48 hours, not clinically significant | 4 | 5 | 5
  48 hours, clinically significant | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline Values in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs were measured in a semi-supine position after 5 minutes rest. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at 1.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post-dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Millimeters of mercury
  SBP, 1.5 hours | -10.4 (15.19) | -6.1 (11.86) | -3.8 (7.65)
  SBP, 2 hours | -10.3 (10.99) | -7.5 (7.82) | -0.1 (11.96)
  SBP, 4 hours | -6.2 (11.53) | -3.0 (8.85) | 0.5 (9.61)
  SBP, 8 hours | -10.1 (9.64) | -0.5 (8.25) | -2.9 (6.79)
  SBP, 12 hours | -5.1 (9.43) | -0.6 (8.00) | -1.9 (12.78)
  SBP, 24 hours | -9.8 (15.75) | -6.6 (11.58) | -4.9 (8.10)
  SBP, 36 hours | -7.3 (13.98) | 2.0 (8.86) | -2.6 (12.64)
  SBP, 48 hours | -6.7 (13.08) | -10.6 (19.38) | -5.3 (14.04)
  DBP, 1.5 hours | -6.8 (8.84) | -3.5 (7.05) | 1.1 (9.25)
  DBP, 2 hours | -6.4 (6.13) | -5.1 (6.29) | 2.4 (7.17)
  DBP, 4 hours | -3.8 (7.12) | -0.9 (6.75) | 3.4 (6.19)
  DBP, 8 hours | -7.0 (4.80) | -2.9 (5.51) | -0.8 (7.69)
  DBP, 12 hours | -5.4 (3.64) | -3.1 (6.24) | 1.9 (7.26)
  DBP, 24 hours | -8.4 (8.69) | -3.4 (12.00) | -1.0 (10.68)
  DBP, 36 hours | -9.3 (7.26) | -1.3 (5.50) | -1.1 (6.33)
  DBP, 48 hours | -6.6 (8.38) | 0.9 (11.32) | 0.8 (6.18)

12. Secondary Outcome: Change From Baseline Values in Heart Rate
Description: Vital signs was measured in a semi-supine position after 5 minutes rest. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1) and at 1.5 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, and 48 hours post dose
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Beats per minute
  1.5 hours | 0.3 (7.47) | 0.6 (9.86) | -0.6 (6.50)
  2 hours | -0.8 (7.98) | -0.1 (10.20) | 0.8 (5.60)
  4 hours | -3.7 (8.79) | 1.4 (4.44) | 0.1 (6.77)
  8 hours | -1.3 (7.91) | 2.6 (4.90) | 1.0 (4.93)
  12 hours | 3.9 (12.23) | 4.8 (3.58) | 5.1 (7.26)
  24 hours | -4.3 (6.78) | -1.1 (6.64) | -2.0 (8.12)
  36 hours | 3.8 (9.76) | 3.8 (3.20) | 2.4 (9.68)
  48 hours | -0.7 (3.94) | 2.8 (7.19) | -0.9 (6.56)

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgment.
Time Frame: Up to Day 15
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Participants
  Any Non-SAE | 3 | 2 | 4
  Any SAE | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Toxicity Grading 3 or Higher for Clinical Chemistry Parameters
Description: Blood samples were collected to measure the number of participants with toxicity grades higher than 3 or 4, for urea, Creatine kinase (CK), creatinine, glucose, sodium, potassium, calcium, Aspartate Aminotransferase, (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) levels, total and direct bilirubin, total protein, and albumin.
Time Frame: Up to Day 15
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Participants | 0 | 1 | 6

15. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: ALT, ALP, AST and CK
Description: Blood samples were collected to analyze clinical chemistry parameters including: ALT, ALP, AST and CK. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Day 2
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 6
International units per liter
  ALT, Day 2 | -2.1 (5.90) | -0.1 (4.19) | -3.7 (6.59)
  ALP, Day 2 | -1.3 (7.98) | -4.4 (5.21) | -5.2 (4.36)
  AST, Day 2 | -1.8 (2.59) | -1.5 (4.31) | -7.8 (10.59)
  CK, Day 2 | -52.9 (57.31) | -36.4 (35.73) | -32.3 (79.05)

16. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected to analyze clinical chemistry parameters including albumin and protein. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Day 2
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 6
Grams per liter
  Albumin, Day 2 | -1.3 (2.35) | -0.4 (1.60) | -1.7 (2.80)
  Protein, Day 2 | -0.9 (4.26) | 0.8 (2.82) | -3.5 (5.72)

17. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected to analyze clinical chemistry parameters including bilirubin, direct bilirubin and creatinine. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Day 2
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 6
Micromoles per liter
  Bilirubin, Day 2 | -2.470 (4.6131) | -1.924 (4.9592) | -7.695 (12.6932)
  Creatinine, Day 2 | -3.2413 (5.97927) | 7.6245 (15.89752) | -0.4420 (4.83379)
  Direct bilirubin, Day 2 | -0.3230 (0.71250) | -0.5771 (0.89060) | -1.8525 (2.71759)

18. Secondary Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Urea
Description: Blood samples were collected to analyze clinical chemistry parameters including calcium, glucose, potassium, sodium and urea. Baseline is defined as Day 1 (Pre-Dose). Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline and at Day 2
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 6
Millimoles per liter
  Calcium, Day 2 | -0.00831 (0.065033) | -0.01623 (0.059119) | -0.05488 (0.092641)
  Glucose, Day 2 | -0.08016 (0.514103) | 0.04855 (0.755546) | -0.79563 (2.183639)
  Potassium, Day 2 | 0.01 (0.481) | 0.35 (0.307) | 0.02 (0.337)
  Sodium, Day 2 | -0.4 (1.67) | 0.6 (2.33) | 0.7 (1.97)
  Urea, Day 2 | 0.1983 (0.92942) | 0.4909 (1.29336) | 0.2975 (0.57194)

19. Secondary Outcome: Number of Participants With Toxicity Grading 3 or Higher for Hematology Parameters
Description: Blood samples were collected to measure the number of participants with toxicity grades higher than 3 or 4 for blood neurtophils and blood platelets.
Time Frame: Up to 15 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Participants | 0 | 0 | 2

20. Secondary Outcome: Number of Participants With Toxicity Grading 3 or Higher for Urinalysis Parameters
Description: Urine samples were collected and specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones were analyzed by dipstick method.
Time Frame: Up to 15 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Participants | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Abnormal Findings During Physical Examinations
Description: A complete physical examination included, at a minimum, assessments of the skin, cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight were also measured and recorded. A brief physical examination included, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Pre-dose up to 31 days prior to dosing
Population: Safety Population. This analysis was planned but data was not captured in the database.
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Total Unchanged Drug (Ae_total) and Amount of Drug Excreted in Urine in a Time Intervals (Ae (t1-t2) for Gepotidacin
Description: Urine samples were collected from participants at indicated time points. Ae_total was calculated by adding all the fractions of drug collected over all the allotted time intervals. Ae (t1-t2) was the amount of drug excreted in urine in time intervals for predose, 0 to 6, 6 to 12, 12 to 24, 24 to 36, and 36 to 48 hours after dosing for participants with hepatic impairment; and predose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours for participants with normal hepatic function. It was calculated by multiplication of the urine concentration for a time interval and the length of this time interval.
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 8 | 8
Milligrams
  Ae_total, n=6, 6, 6: number analyzed (Participants) | 6 | 6 | 6
  Ae_total, n=6, 6, 6 | 127.67 (63.552) | 191.39 (84.368) | 325.31 (124.273)
  Ae (0-2), n=8, 0, 0: number analyzed (Participants) | 8 | 0 | 0
  Ae (0-2), n=8, 0, 0 | 5.82 (7.838) |  |
  Ae (2-4), n=9, 0, 0: number analyzed (Participants) | 9 | 0 | 0
  Ae (2-4), n=9, 0, 0 | 55.53 (55.735) |  |
  Ae (4-6), n=9, 0, 0: number analyzed (Participants) | 9 | 0 | 0
  Ae (4-6), n=9, 0, 0 | 28.79 (19.702) |  |
  Ae (0-6), n=0, 7, 8: number analyzed (Participants) | 0 | 7 | 8
  Ae (0-6), n=0, 7, 8 |  | 144.24 (104.112) | 199.28 (103.407)
  Ae (6-8), n=9, 0, 0: number analyzed (Participants) | 9 | 0 | 0
  Ae (6-8), n=9, 0, 0 | 18.67 (8.371) |  |
  Ae (6-12), n=0, 7, 8: number analyzed (Participants) | 0 | 7 | 8
  Ae (6-12), n=0, 7, 8 |  | 60.53 (35.231) | 112.65 (93.439)
  Ae (8-12), n=9, 0, 0: number analyzed (Participants) | 9 | 0 | 0
  Ae (8-12), n=9, 0, 0 | 16.21 (7.056) |  |
  Ae (12-24), n=7, 6, 7: number analyzed (Participants) | 7 | 6 | 7
  Ae (12-24), n=7, 6, 7 | 11.15 (6.007) | 12.72 (7.265) | 23.27 (17.258)
  Ae (24-36), n=8, 7, 7: number analyzed (Participants) | 8 | 7 | 7
  Ae (24-36), n=8, 7, 7 | 6.62 (4.675) | 8.44 (3.914) | 12.78 (6.869)
  Ae (36-48), n=6, 8, 7: number analyzed (Participants) | 6 | 8 | 7
  Ae (36-48), n=6, 8, 7 | 3.71 (1.845) | 4.59 (3.512) | 6.04 (2.909)

23. Secondary Outcome: Percentage of the Given Dose of Drug Excreted in Urine (Fe%)
Description: Urine samples were collected from participants at indicated time points. Percentage of the given dose of drug excreted in urine was calculated as: (Ae_total divided by Dose) and multiplied by 100.
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of drug
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6
Percentage of drug | 8.51 (4.237) | 12.76 (5.625) | 21.69 (8.285)

24. Secondary Outcome: Renal Clearance (CLr) of Gepotidacin
Description: Urine samples were collected from participants at indicated time points. Renal clearance for gepotidacin was calculated as Ae_total divided by AUC (0-t).
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 6
Liters per hour | 8.18 (3.209) | 9.45 (2.710) | 12.46 (3.911)

25. Secondary Outcome: AUC(0-12) of Gepotidacin
Description: Urine samples were collected from participants at indicated time points to evaluate AUC(0-12) PK parameter of gepotidacin.
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours and 8-12 hours post dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 9 | 7 | 8
Hours*micrograms per milliliter | 1201 (1033.5) | 3030 (2245.5) | 4771 (4678.3)

26. Secondary Outcome: AUC(0-24) of Gepotidacin
Description: Urine samples were collected from participants at indicated time points to evaluate AUC(0-24) PK parameter of gepotidacin.
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-12 hours and 12-24 hours post dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 6 | 7
Hours*micrograms per milliliter | 1269 (1040.4) | 2925 (1868.3) | 5807 (5151.0)

27. Secondary Outcome: AUC(0-48) of Gepotidacin
Description: Urine samples were collected from participants at indicated time points to evaluate AUC(0-48) PK parameter of gepotidacin.
Time Frame: Pre-dose, 0-2 hours, 2-4 hours, 4-6 hours, 6-8 hours, 8-12 hours, 12-24 hours, 24-36 hours and 36-48 hours post dose
Population: PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 5 | 6
Hours*micrograms per milliliter | 1394 (1252.4) | 3547 (1667.9) | 5035 (4695.6)

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the treatment up to 15 days
Description: Non-serious AEs and SAEs were collected for Safety population
Arm/Group | Participants With Normal Hepatic Function | Participants With Moderate Hepatic Impairment | Participants With Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/9 | 2/8 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Normal Hepatic Function (N=9) | Participants With Moderate Hepatic Impairment (N=8) | Participants With Severe Hepatic Impairment (N=8)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Normal Hepatic Function (N=9) | Participants With Moderate Hepatic Impairment (N=8) | Participants With Severe Hepatic Impairment (N=8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03562117/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03562117/SAP_001.pdf